CLINICAL TRIAL: NCT02214316
Title: IVF in Pediatric Concussion
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201408006
Record Dates: First submitted 2014-08-07; First posted 2014-08-12 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Pediatric Mild Traumatic Brain Injury
MeSH Terms: interventions — Saline Solution, Hypertonic

ARMS (1):
- Interventional 1 (Experimental): Interventional experimental arm with hypertonic saline
  Interventions: Other: Hypertonic Saline

INTERVENTIONS:
Other: Hypertonic Saline

SUMMARY:
Children with concussion may improve with intravenous fluids.

ELIGIBILITY:
Inclusion Criteria:

* History of acute concussion

Exclusion Criteria:

* Other significant medical illness

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Postconcussive symptoms | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States